CLINICAL TRIAL: NCT01163695
Title: The SUUBI Program: Creating Asset-Ownership Opportunities and Health Promotion Among Orphaned Children in Uganda
Brief Title: The SUUBI Program: Asset-Ownership for Orphaned Children in Uganda
Acronym: SUUBI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Fred Ssewamala, PhD, Associate Professor of Social Work, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAA5337; R21MH076475-01 (NIH)
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Poverty
Keywords: economic empowerment model, orphans, sub-Saharan Africa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Children's development account — Children in the experimental condition (the SUUBI program) received, in addition to the usual care, an economic empowerment intervention aimed at promoting asset accumulation for families-and consisting of three major components: 1) workshops focused on asset-building and future planning; 2) a monthly mentorship program for adolescents with peer mentors on life options; and 3) a Child Development Account (CDA), dedicated to paying for secondary schooling, vocational training and/or a family small business. The CDAs were matched savings accounts, with a match rate of 2:1 as an incentive for participants to save, but with a limit on the maximum savings that could be matched (the match cap, in this case, was equivalent to $10 a month).
  Other Names: Children's savings account

SUMMARY:
This study examines an economic empowerment model of care and support for orphaned adolescents in rural Uganda. The Suubi intervention focuses on economic empowerment of families caring for orphaned youths. It attempts to address the health risks and poor educational achievements resulting from poverty and limited options.

DETAILED DESCRIPTION:
The AIDS epidemic and a 20-year civil war have had a devastating impact on Uganda. The events have led to population displacement, worsening living conditions, exacerbation of poverty, and disruption of already weakened social service systems. As implemented, the Suubi Project goes considerably beyond the usual care, which primarily consists of institutionalization and reactive strategies (involving food and material aid). Specifically, the intervention promotes children's savings accounts, also known as children development accounts, for postprimary education and microenterprise development (i.e., development of small income-generating businesses).

The Suubi intervention is grounded in asset theory (Sherraden 1990, 1991), which holds that assets (e.g., savings, educational opportunities, and economic opportunities in the form of income-generating activities or microenterprises) have important economic, social, and psychological benefits for individuals and families. Asset building is increasingly viewed as a critical factor for reducing poverty, improving psychosocial functioning, and positively affecting attitudes and behaviors.

ELIGIBILITY:
Inclusion Criteria:

* an orphaned child, defined as a child who has lost one or both parents to HIV/AIDS; enrolled in primary school (even though possibly not attending regularly); between the ages of 12 to 15 years.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 286 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Savings and asset-accumulation | baseline, 10-month and 20-month post-intervention
  past experience, current savings, and attitudes toward saving

SECONDARY OUTCOMES:
Sexual risk taking | baseline, 10-month and 20-month post-intervention
  Sexual risk taking behavior (history and onset of sexual intercourse), Intentions to engage in sexual risk behaviors
Educational outcomes | baseline, 10-month, and 20-month post-intervention
  School enrollment, School attendance, School grades, Educational aspirations
Mental health | baseline, 10-month and 20-month post-intervention
  Self-esteem, depression, hopelessness, helplessness
Social and family support | baseline, 10-month and 20-month post-intervention
  Emotional support from caregivers, practical assistance, financial assistance and advice/guidance, and family communication

CONTACTS AND LOCATIONS:
Overall Officials: Fred M Ssewamala, PhD, Principal Investigator — Columbia University
Locations (1):
- St. Joseph's Matale Parish, Rakai, Rakai, Uganda

REFERENCES:
- [Result] Ssewamala FM, Ismayilova L, McKay M, Sperber E, Bannon W Jr, Alicea S. Gender and the effects of an economic empowerment program on attitudes toward sexual risk-taking among AIDS-orphaned adolescent youth in Uganda. J Adolesc Health. 2010 Apr;46(4):372-8. doi: 10.1016/j.jadohealth.2009.08.010. PMID 20307827
- [Result] Ssewamala FM, Han CK, Neilands TB, Ismayilova L, Sperber E. Effect of economic assets on sexual risk-taking intentions among orphaned adolescents in Uganda. Am J Public Health. 2010 Mar;100(3):483-8. doi: 10.2105/AJPH.2008.158840. Epub 2010 Jan 14. PMID 20075323
- [Result] Ssewamala FM, Han CK, Neilands TB. Asset ownership and health and mental health functioning among AIDS-orphaned adolescents: findings from a randomized clinical trial in rural Uganda. Soc Sci Med. 2009 Jul;69(2):191-8. doi: 10.1016/j.socscimed.2009.05.019. Epub 2009 Jun 10. PMID 19520472
- [Result] Ssewamala FM, Alicea S, Bannon WM Jr, Ismayilova L. A novel economic intervention to reduce HIV risks among school-going AIDS orphans in rural Uganda. J Adolesc Health. 2008 Jan;42(1):102-4. doi: 10.1016/j.jadohealth.2007.08.011. PMID 18155037
- [Derived] Ismayilova L, Ssewamala FM, Karimli L. Family support as a mediator of change in sexual risk-taking attitudes among orphaned adolescents in rural Uganda. J Adolesc Health. 2012 Mar;50(3):228-35. doi: 10.1016/j.jadohealth.2011.06.008. Epub 2011 Aug 27. PMID 22325127